CLINICAL TRIAL: NCT01769105
Title: Prospective, Randomized, Controlled Comparison of an Automated Thermal Pulsation Treatment (Lipiflow ®) and a Standard Lid Hygiene Regime
Brief Title: Comparison of Lipiflow®-Treatment and a Standard Lid Hygiene Regime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, David Finis, MD, Principal investigator, department of ophthalmology, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HHUAU052012
Record Dates: First submitted 2013-01-11; First posted 2013-01-16 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian Gland Dysfunction; Lipiflow
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Lid Hygiene Regime (Active Comparator): Patients receive detailed verbal and written instruction to perform lid hygiene twice daily
  Interventions: Behavioral: Lid hygiene regime
- Lipiflow (Active Comparator): Patients receive a singe Lipiflow-treatment
  Interventions: Device: Lipiflow

INTERVENTIONS:
Device: Lipiflow — Patients receive a single Lipiflow-treatment
  Arms: Lipiflow
Behavioral: Lid hygiene regime — Patients receive verbal and written instruction to perform lid hygiene twice daily
  Arms: Standard Lid Hygiene Regime

SUMMARY:
Recently, beneficial effects on Meibomian gland dysfunction (MGD) of a single automated thermal pulsation with the Lipiflow® system have been reported in several case reports. In one study this treatment was compared with hyperthermia (iheat®) for 4 weeks. However, treatment recommendations for lid hygiene according to the MGD-report consist of hyperthermia followed by lid massage and lid margin cleansing over several months. To the best of the investigators knowledge this is the first randomized prospective study to compare automated thermal pulsation treatment with the new Lipiflow ® system with a standard lid hygiene regime.

The investigators suggest that a single treatment with Lipiflow® is superior to a lid hygiene regime.

DETAILED DESCRIPTION:
Once a patient has been identified as a possible candidate for the study, he/she is first informed verbally and in writing about the study. After signing the consent form he/she will be randomized to either the Lipiflow® treatment (Lipiflow® group) or alternatively be given an instruction sheet and a verbal explanation for lid warming and massage (lid hygiene group). After 3 month a cross-over of the lid hygiene group to the Lipiflow® group is conducted.

A full examination is performed before and 4 weeks and 3 months after therapy. All tests are performed by a physician or trained graduate students of the Department of Ophthalmology, Heinrich-Heine University. The examiner is blinded, i.e. he does not know which treatment the patient will receive or receiving.

Treatment Lipiflow®:

The automated thermal pulsation with Lipiflow® provides is a low risk therapy. After local anesthesia the applicators are inserted. These look like a kind of goggles and consist of two parts which embrace the eyelids from the front and from behind. Through the rear part heat is applied to a maximum of 42.5° C. By isolating the heat remains on the eyelid limited. Through the front part the gland a massage is performed. The treatment takes 12 minutes per eye and can be done depending on the patient's wishes simultaneously or one eye after the other. The therapy is approved by the FDA as a medical technical innovation and has also been approved by ISO and CE Mark certification for use in Europe. Irritation or minor trauma of the eyelids and the conjunctiva and cornea, as well as a violation of the eyelids and the conjunctiva and cornea are theoretically possible, but extremely unlikely. Permanent damages to the eyes have not been reported in the literature.

In the unlikely event, that complications occur during treatment, requiring an additional treatment, this is performed in the department of ophthalmology of the Heinrich-Heine University Duesseldorf.

Test parameters:

At any time of investigation, the following parameters are evaluated:

Lipiview®, Tear Lab®, Schirmer test, break-up time, corneal and conjunctival fluorescein staining, Meibomian gland evaluation (MGE), examination of the eyelids, Meibography, OSDI score, SPEED score

All test parameters are established procedures and have in common a very low risk of harm to the patient. In detail:

The Lipiview® is a device that quantifies the thickness of the lipid layer of the tear film using interferometry. For this the patient looks into a kind of camera while recordings of his tear film are made, which are then analyzed by a computer.

Tear Lab® is a method for measuring tear film osmolarity. A pen-like instrument (the osmometer) is held on the tear meniscus and collects 100 nl tears within fractions of a second in the unit. There is no need for local anaesthesia. By electrical impedance measurement, then the tear film osmolarity is measured. The examiner can then read the values digitally.

The Schirmer test consists of a strip of filter paper that is placed in the conjunctival sac of the patient for five minutes. The filter paper absorbs the tear fluid and the stained by the tear fluid line serves as a measure of tear secretion.

Tear break-up time is the time between a blink and the tear film shows signs of breaking up. In this study this is measured non-invasive with the Oculus-Keratograph 5 M®. The patient looks into a kind of camera while recordings of his tear film are made which are then analyzed by a computer.

Vital corneal and conjunctival epithelium cannot be stained by fluorescein. The dye adheres to nonviable cells. The degree of staining, can be judged by the investigator by slit-lamp examination.

For evaluation of the secreting meibomian glands a specialized device (Meibomian gland evaluator) is used, that provides a defined pressure to the lid. The examiner observes the ducts of the Meibomian glands and assesses how many glands are yielding secretion.

Examination of the eyelids is done using a slit lamp to assess a thickening or a significant vascularisation the lid margin.

To perform meibography the lids are illuminated by infrared light. Functional acini of the glands become clearly visible and can be differentiated from atrophic acini. The number of atrophic meibomian glands can be counted by a score.

OSDI (Ocular-Surface-Disease-Index) and SPEED (Standard Pattern Evaluation of Eye Dryness) are questionnaires to quantify the symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* All patients with meibomian gland dysfunction requiring treatment (defined below),
* who have given their written consent to the study.
* Meibomian gland dysfunction requiring treatment is classified by us as:
* Speed score> 7, Lipiview <61 nm, MGE <5 of 15 open glands

Exclusion Criteria:

* Excluded are patients who, due to other diseases would not be able to fulfill the follow-up appointments or give an informed consent to the study
* Systemic medication with tetracyclin derivatives, antihistamines, isotretinoin, or nutritional supplements for MGD that started <3 months before baseline examination
* Topical cyclosporine-A or steroids that started <1 month before baseline examination
* Ocular surgery or trauma <3 months before baseline examination
* Any eyelid abnormalities
* Systemic diseases resulting in dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Geerling, M.D., Study Chair — Deparmtent of ophthalmology, Heinrich-Heine-University, Duesseldorf
Locations (1):
- Deparment of ophthalmology, Heinrich-Heine-University, Düsseldorf, Germany

REFERENCES:
- [Result] Finis D, Hayajneh J, Konig C, Borrelli M, Schrader S, Geerling G. Evaluation of an automated thermodynamic treatment (LipiFlow(R)) system for meibomian gland dysfunction: a prospective, randomized, observer-masked trial. Ocul Surf. 2014 Apr;12(2):146-54. doi: 10.1016/j.jtos.2013.12.001. Epub 2014 Jan 22. PMID 24725326

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five patients had been enrolled in the study, but withdrew their participation after baseline examination for personal reasons. They did not receive any treatment.
Groups:
- Standard Lid Hygiene Regime First, Then Lipiflow: Patients receive detailed verbal and written instruction to perform lid hygiene twice daily, then Lipiflow
  Lid hygiene regime: Patients receive verbal and written instruction to perform lid hygiene twice daily and after 3 month a single Lipiflow treatment
Period: First Intervention
Arm/Group | Standard Lid Hygiene Regime First, Then Lipiflow | Lipiflow
Started | 16 | 19
Completed | 14 | 17
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 2
Period: Cross-over
Arm/Group | Standard Lid Hygiene Regime First, Then Lipiflow | Lipiflow
Started | 14 | 0 (Cross-over was only intended for the Lid margin hygiene group)
Completed | 9 | 0 (Was not intended by the study protocol)
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Lid Hygiene Regime First, Then Lipiflow: Patients receive detailed verbal and written instruction to perform lid hygiene twice daily, then Lipiflow
  Lid hygiene regime: Patients receive verbal and written instruction to perform lid hygiene twice daily, then a single Lipiflow-treatment
- Total: Total of all reporting groups
Arm/Group | Standard Lid Hygiene Regime First, Then Lipiflow | Lipiflow | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (19) | 45 (23) | 47 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Germany | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change of Dry Eye Symptoms
Description: The symptoms of dry eyes are measured in our study with the OSDI and the SPEED questionaire. Primary outcome measure (OSDI)
  Patients completed two symptom questionnaires: OSDI (Ocular Surface Disease Index) and SPEED (Standard Patient Evaluation of Eye dryness).
  OSDI scores range from 0 (no symptoms) to 100 (severe symptoms). SPEED scores range from 0 (no symptoms) to 28 (severe symptoms). So a reduction of the OSDI or SPEED score indicates an improvement of subjective dry eye symptoms.
Time Frame: after 3 month compared to baseline value
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cross-over Lipiflow: patients received a single Lipiflow treatment after performing lid hygiene for 3 month
Arm/Group | Standard Lid Hygiene Regime | Lipiflow | Cross-over Lipiflow
Number analyzed (Participants) | 14 | 17 | 9
units on a scale
  OSDI Baseline | 40.1 (16.7) | 46.2 (14.8) | 39.7 (23.6)
  SPEED Baseline | 15.9 (6.6) | 16.8 (5.6) | 14.7 (7.7)
  OSDI 3 month | 40.0 (23.4) | 34.6 (19.6) | 32.8 (24.4)
  SPEED 3 month | 14.7 (7.1) | 14.5 (7.2) | 12.6 (6.5)

2. Secondary Outcome: Change of Break-up-time
Description: break-up-time is measured non-invasive with the Oculus Keratograph 5 M;
  The break-up-time is measured in seconds. A low break-up-time suggests a lower lipid layer thickness. A higher break-up-time can be regarded as an improvement of ocular surface lubrication.
Time Frame: after 3 month compared to baseline value
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Cross-over Lipiflow: Patients receive Lipiflow after performing Lid hygiene for 3 month
Arm/Group | Standard Lid Hygiene Regime | Lipiflow | Cross-over Lipiflow
Number analyzed (Participants) | 14 | 17 | 9
seconds
  Baseline | 7.7 (6.1) | 7.9 (8.5) | 6.7 (6.1)
  After 3 month | 7.5 (6.1) | 9.9 (7.0) | 7.3 (5.1)

3. Secondary Outcome: Change in Tear Film Osmolarity
Description: osmolarity is measured with the tear-lab;
  The osmolarity is measured in mOsm/l. A higher osmolarity can be regarded as an objective sign of dry eye disease.
  A lower osmolarity after therapy can be regarded as an improvement of ocular surface disease.
Time Frame: after 3 month compared to baseline value
Measure: Mean (Standard Deviation); unit: mOsm/L
Arm/Group | Standard Lid Hygiene Regime | Lipiflow | Cross-over Lipiflow
Number analyzed (Participants) | 14 | 17 | 9
mOsm/L
  Baseline | 296.7 (10.2) | 301.5 (11.4) | 305.0 (8.7)
  After 3 month | 303.7 (8.1) | 307.1 (14.0) | 310.0 (7.4)

4. Secondary Outcome: Change in Lipid Layer Thickness
Description: lipid layer thickness (LLT) is measured with the Lipiview-interferometer;
  High values of LLT indicate a better lubrication of the ocular surface, so an increase in LLT can be regarded in an improvement of ocular surface.
  LLT is measured in Interferometric color units (ICUs) whereas 1 ICU reflects about 1 nm lipid layer thickness.
Time Frame: after 3 month compared to baseline value
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Standard Lid Hygiene Regime | Lipiflow | Cross-over Lipiflow
Number analyzed (Participants) | 14 | 17 | 9
nm
  Baseline | 44.1 (7.9) | 43.4 (9.9) | 45.8 (21.8)
  After 3 month | 46.4 (20.8) | 47.4 (16.7) | 59.2 (26.3)

5. Secondary Outcome: Change in Expressible Meibomian Glands
Description: expressible Meibomian glands are measured with the Meibomian gland evaluator; A higher number of expressible Meibomian glands indicate a lower likelihood Meibomian Gland dysfunction.
Time Frame: after 3 month compared to baseline value
Measure: Mean (Standard Deviation); unit: number of expressible glands
Arm/Group | Standard Lid Hygiene Regime | Lipiflow | Cross-over Lipiflow
Number analyzed (Participants) | 14 | 17 | 9
number of expressible glands
  Baseline | 2.1 (1.3) | 2.5 (1.4) | 4.1 (2.5)
  After 3 month | 4.6 (3.8) | 5.5 (3.6) | 5.8 (3.2)

ADVERSE EVENTS:
Time Frame: 3 month
Groups:
- Standard Lid Hygiene Regime First, Then Lipiflow: Patients receive detailed verbal and written instruction to perform lid hygiene twice daily first and then Lipiflow
  Lid hygiene regime: Patients receive verbal and written instruction to perform lid hygiene twice daily and after 3 month a single Lipiflow-treatment
Arm/Group | Standard Lid Hygiene Regime First, Then Lipiflow | Lipiflow
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

LIMITATIONS AND CAVEATS:
For further information please have a look at Finis et al: Evaluation of an automated thermodynamic treatment (LipiFlow®) system for meibomian gland dysfunction: a prospective, randomized, observer-masked trial.Ocul Surf. 2014 Apr;12(2):146-54.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes